CLINICAL TRIAL: NCT04839068
Title: The Impact of COVID -19 Pandemic Stress on Sex Ratio at Birth and Other Pregnancy Outcomes
Brief Title: the Impact of Covid-19 Pandemic Stress on Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Ahmed Abdelreheem, Principal investigator, Assiut University
Other Study IDs: covid2021
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First is retrospective part: : by obtaining the data from the patients records in a period between January 1st 2019 to December 31st 2019, and from May 1st 2020 to December (excluding women conceived before April 1st 2020)
  Interventions: Device: covid 19 on pregnancy outcomes
- Second is prospective part: the same data will be obtained from the patient records in the same way in a period from the January 1st 2021 to the December 31st to assess the pregnancy outcomes in pregnant women who conceived after occurrence of Covid 19 pandemic in Egypt.
  Interventions: Device: covid 19 on pregnancy outcomes

INTERVENTIONS:
Device: covid 19 on pregnancy outcomes — covid 19 on pregnancy outcomes and sex ratio at birth

SUMMARY:
This study is aiming to evaluate the effects of the COVID-19 pandemic stress on pregnancy outcomes including the sex ratio at birth.

DETAILED DESCRIPTION:
* Coronavirus disease 2019 (COVID-19) is an emerging respiratory disease caused by a single-strand, positive-sense ribonucleic acid (RNA) virus, severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) virus (Masters, 2019).
* The sex ratio (ratio of boys to girls) at birth (SRB) is about 1.01-1.05 in most populations (Abdoli, 2020). Various influencing factors affect the SRB, including maternal stress, endocrine disruption, maternal inflammatory responses and maternal nutrition (Lipner et al., 2019).
* These stressful life events consequently influence on maternal immunological and endocrine conditions, and the male fetuses are more vulnerable to be affected by these conditions. It is of interest that male fetus is biologically weaker and more susceptible to prenatal events and diseases than female fetuses. Hence, premature death is higher in boys than girls (Ahrenfeldt et al., 2017).
* The recent pandemic of the coronavirus disease 2019 (COVID-19) has been known to have various impacts on pregnant women (Rasmussen et al., 2020). Placentas of infected mothers show inflammatory, vascular and thrombotic changes (Prochaska et al., 2020). Among the neonates, children and adults (Bjelosevic et al., 2017), higher morbidity and mortality of males than females were reported. It is observed that the incidence of stillbirth was significantly increased during the pandemic period than during the pre pandemic period in London, UK (Khalilet al., 2020).
* The start of appearance of Covid 19 cases in Egypt was in March 2020, with subsequent increase in cases with its peak in May, June and July 2020, with lockdown and social and financial affection with great stress on families

ELIGIBILITY:
Inclusion Criteria:

- 1. All pregnant women attended to the Women health hospital in a period from January 1st 2019 to December 31st 2019 for child birth or miscarriage (either first or second trimesters) or ectopic or molar pregnancies.

2. All pregnant women attended to the Women health hospital in a period from May 1st 2020 to December 31st 2021 for child birth or miscarriage (either first or second trimesters) or ectopic or molar pregnancies management.

Exclusion Criteria:

* 3. Pregnant women attended to the Women health hospital in a period from April 1st 2020 to December 31st 2021 for child birth or miscarriage (either first or second trimesters) or ectopic or molar pregnancies management who conceived before April 1st 2020

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: c. Sample Size Calculation: As our study is a descriptive study aiming to explore the changes in sex ratios and other pregnancy outcomes in different months of the two years before and after COVID-19 pandemic. We will include all eligible records during those years (total coverage sample). Expected number per year according to previous records is 7000 cases
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The effect of Covid 19 pandemic stress on sex ratio at birth | one year

CONTACTS AND LOCATIONS:
Locations (1):
- The Clinical Obstetrics and Gynaecology department, Assuit University Hospital, Egypt, Asyut, Egypt